CLINICAL TRIAL: NCT02456636
Title: Rural Engagement in Primary Care for Optimizing Weight Reduction (RE-POWER)
Brief Title: Rural Engagement in Primary Care for Optimizing Weight Reduction
Acronym: RE-POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE-POWER; PCORI-1402-09413 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute); STUDY00002654 (Other: KUMC IRB)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Obesity
Keywords: Weight loss; Weight management; Diabetes; Heart disease
MeSH Terms: conditions — Obesity; Weight Loss; Diabetes Mellitus; Heart Diseases | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fee-for-Service Model (FFS, In clinic individual visits) (Active Comparator): Participants will receive individual counseling from their physician or other healthcare professional during regular clinic visits.
  Interventions: Behavioral: Fee-for-Service Model (FFS, In clinic individual visits)
- Patient Centered Medical Home (PCMH, In clinic group visits) (Active Comparator): Participants will take part in group weight-management counseling during in-person group visits; later sessions may be conducted via group telephone calls if the group prefers.
  Interventions: Behavioral: Patient Centered Medical Home (PCMH, In clinic group visits)
- Disease Management (DM, Phone group visits) (Active Comparator): Participants will take part in group weight-management counseling by telephone.
  Interventions: Behavioral: Disease Management (DM, Phone group visits)

INTERVENTIONS:
Behavioral: Fee-for-Service Model (FFS, In clinic individual visits) — To be performed by participant's doctor or other healthcare professional in their doctor's office.
  Other Names: Individual weight management counseling
  Arms: Fee-for-Service Model (FFS, In clinic individual visits)
Behavioral: Patient Centered Medical Home (PCMH, In clinic group visits) — To be performed by a registered dietitian, a nurse or other healthcare professional in their local setting.
  Other Names: Group weight management counseling (in-person and telephone)
  Arms: Patient Centered Medical Home (PCMH, In clinic group visits)
Behavioral: Disease Management (DM, Phone group visits) — To be performed by obesity treatment specialists with relevant graduate training and experience with weight loss counseling via telephone.
  Other Names: Group weight management counseling (telephone)
  Arms: Disease Management (DM, Phone group visits)

SUMMARY:
The purpose of this study is to compare three methods for managing obesity in rural patients, to see which method will result in patients being able to attain their weight loss goal and maintain that weight loss.

DETAILED DESCRIPTION:
Nearly 20% of the U.S. population lives in rural communities. Rural residents suffer at a higher rate from obesity and obesity-related illnesses, including diabetes, heart disease, and arthritis. Local primary care physicians are an important resource for treating obesity in rural areas because of a lack of other community resources.

This study is looking at how effective current, real-world primary care treatment models are in helping rural residents lose weight and maintain that weight loss. Physician clinics will be randomized (like picking numbers from a hat) to conduct one of the three methods. The method a participant is part of will depend on the method their physician's clinic is randomized to. The three methods involved in this study are:

1. Individual weight-management counseling in person (in clinic individual visits)
2. Group weight-management counseling, both in person and by telephone; the latter if preferred by the group (in clinic group visits)
3. Group weight-management counseling by telephone (phone group visits)

Participants will be in the study about 24 months. The number of in-person clinic visits and phone calls each participant will be asked to complete depends on the method.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 kg/m2 and 45 kg/m2.
* Live in a rural location.
* Have clearance from their primary care provider to participate in a diet and exercise weight control intervention.
* Have access to a telephone.
* One individual per household will be permitted to enroll in the study.

Exclusion Criteria:

* History of heart attack in the last six months, stroke in the last six months, or new cancer diagnosis in the last six months.
* History of bariatric surgery or planning bariatric surgery in the next two years.
* Pregnancy within the last six months or planned within the next two years or currently pregnant or lactating.
* Serious medical conditions where weight loss is contraindicated.
* End stage renal disease or end stage liver disease.
* Other medical contraindications as determined by the patient's primary care physician (PCP); documented PCP clearance will be obtained.
* Participants who are already enrolled in, or planning to enroll in another research study where weight loss is targeted.
* Participants who plan to relocate outside of their provider's service area or who plan to leave their primary care clinic in the next 2 years.
* Unable to read and understand English.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1432 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christie Befort, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Saint Onge JM, Fagan M, Befort CA. The association between the obesogenic environment and 6-month and 24-month weight change in a rural weight loss intervention trial in the United States. Prev Med. 2022 May;158:107040. doi: 10.1016/j.ypmed.2022.107040. Epub 2022 Apr 7. PMID 35398370
- [Derived] Tang F, Befort CA, Wick J, Gajewski BJ. Unifying the analysis of continuous and categorical measures of weight loss and incorporating group effect: a secondary re-analysis of a large cluster randomized clinical trial using Bayesian approach. BMC Med Res Methodol. 2022 Jan 26;22(1):28. doi: 10.1186/s12874-021-01499-0. PMID 35081912
- [Derived] Katzmarzyk PT, Apolzan JW, Gajewski B, Johnson WD, Martin CK, Newton RL Jr, Perri MG, VanWormer JJ, Befort CA. Weight loss in primary care: A pooled analysis of two pragmatic cluster-randomized trials. Obesity (Silver Spring). 2021 Dec;29(12):2044-2054. doi: 10.1002/oby.23292. Epub 2021 Oct 29. PMID 34714976
- [Derived] Goessl CL, VanWormer JJ, Pathak RD, Ellerbeck EF, Befort CA. Affective disorders, weight change, and patient engagement in a rural behavioral weight loss trial. Prev Med. 2021 Nov;152(Pt 2):106698. doi: 10.1016/j.ypmed.2021.106698. Epub 2021 Jun 24. PMID 34175347
- [Derived] Befort CA, VanWormer JJ, Desouza C, Ellerbeck EF, Gajewski B, Kimminau KS, Greiner KA, Perri MG, Brown AR, Pathak RD, Huang TT, Eiland L, Drincic A. Effect of Behavioral Therapy With In-Clinic or Telephone Group Visits vs In-Clinic Individual Visits on Weight Loss Among Patients With Obesity in Rural Clinical Practice: A Randomized Clinical Trial. JAMA. 2021 Jan 26;325(4):363-372. doi: 10.1001/jama.2020.25855. PMID 33496775
- [Derived] Befort CA, Kurz D, VanWormer JJ, Ellerbeck EF. Recruitment and reach in a pragmatic behavioral weight loss randomized controlled trial: implications for real-world primary care practice. BMC Fam Pract. 2020 Mar 3;21(1):47. doi: 10.1186/s12875-020-01117-w. PMID 32126987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from 36 medical practices were recruited via mailings and in-clinic referrals. Initial eligibility was assessed via telephone screen. Patients then completed a baseline survey, physician clearance was documented, and finally BMI was verified at the initial study visit. The recruitment period was from 2/15/2016 through 10/2/2017.
Groups:
- Fee-for-Service (In Clinic Individual Counseling): Participants will receive individual counseling from their physician or other healthcare professional during regular clinic visits.
  Fee-for-Service Model (FFS): To be performed by participant's doctor or other healthcare professional in their doctor's office.
- Patient Centered Medical Home (In Clinic Group Counseling): Participants will take part in group weight-management counseling during in-person group visits; later sessions may be conducted via group telephone calls if the group prefers.
  Patient Centered Medical Home (PCMH): To be performed by a registered dietitian, a nurse or other healthcare professional.
- Disease Management (Phone Group Counseling): Participants will take part in group weight-management counseling by telephone.
  Disease Management (DM): To be performed by obesity treatment specialists with relevant graduate training and experience with weight loss counseling
Period: Overall Study
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Started | 478 | 479 | 475
6 Month | 474 | 474 | 468
18 Month | 467 | 463 | 461
Completed | 410 | 410 | 400
Not Completed | 68 | 69 | 75
Not completed — Death | 0 | 3 | 0
Not completed — Pregnancy | 1 | 3 | 5
Not completed — Physician Decision | 4 | 5 | 4
Not completed — Withdrawal by Subject | 13 | 14 | 16
Not completed — Lost to Follow-up | 50 | 44 | 50

BASELINE CHARACTERISTICS:
Population: Enrolled minus deaths and medical removals
Groups:
- Total: Total of all reporting groups
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling) | Total
Number analyzed (Participants) | 473 | 468 | 466 | 1407
Age, Categorical [Count of Participants; unit: Participants] — Population: Enrolled minus deaths and medical removals.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 385 | 343 | 372 | 1100
    >=65 years | 88 | 125 | 94 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Enrolled minus deaths and medical removals.
  years | 54.1 (11.5) | 55.7 (12.0) | 54.1 (11.9) | 54.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Enrolled minus deaths and medical removals.
  Participants
    Female | 377 | 343 | 361 | 1081
    Male | 96 | 125 | 105 | 326
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Enrolled minus deaths and medical removals.
  Participants
    White, Non-Hispanic | 463 | 442 | 448 | 1353
    Other | 10 | 26 | 18 | 54
Region of Enrollment [Count of Participants; unit: Participants] — Population: Enrolled minus deaths and medical removals.
  Participants
    United States: Isolated rural | 244 | 203 | 212 | 659
    United States: Small rural | 78 | 83 | 89 | 250
    United States: Large rural | 151 | 182 | 165 | 498
Weight, kg [Mean (Standard Deviation); unit: kg] — Population: Enrolled minus deaths and medical removals
  kg | 103.1 (15.4) | 102.9 (15.5) | 102.7 (15.6) | 102.9 (15.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Enrolled minus deaths and medical removals.
  kg/m^2 | 36.9 (4.0) | 36.7 (3.9) | 36.6 (3.9) | 36.7 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight Change Over 24 Months; Unadjusted Except for Affiliation
Description: Mean weight change (kg) of participants between the three study groups. Weight loss at 24 months, and all relevant study visits in between, will be compared 1) between PCMH (in clinic group visits) versus FFS (in clinic individual visits), 2) between DM (phone group visits) versus FFS (in clinic individual visits), and 3) between PCMH (in clinic group visits) versus DM (phone group visits). Unadjusted except for affiliation.
Time Frame: Baseline and 6, 18 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (97.5% Confidence Interval); unit: kg
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
kg
  Mean Weight change at 6 months | -5.73 [-6.79 to -4.67] | -8.34 [-9.37 to -7.31] | -7.72 [-8.76 to -6.68]
  Mean Weight change at 18 months | -3.35 [-4.57 to -2.14] | -5.58 [-6.77 to -4.39] | -5.17 [-6.37 to -3.97]
  Mean Weight change at 24 months | -2.56 [-3.79 to -1.34] | -4.43 [-5.63 to -3.23] | -3.92 [-5.13 to -2.71]
Statistical Analysis 1: Comparison: Fee-for-Service (In Clinic Individual Counseling) vs Patient Centered Medical Home (In Clinic Group Counseling); PCMH (in clinic group counseling) versus FFS (in clinic individual counseling); Test type: Superiority; p = .025, Mixed Models Analysis; Mean Difference (Net) = -1.87, 97.5% CI 2-sided [-3.51 to -0.23]
Statistical Analysis 2: Comparison: Fee-for-Service (In Clinic Individual Counseling) vs Disease Management (Phone Group Counseling); DM (phone group counseling) versus FFS (in clinic individual counseling); Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = -1.36, 97.5% CI 2-sided [-3.00 to 0.29]
Statistical Analysis 3: Comparison: Patient Centered Medical Home (In Clinic Group Counseling) vs Disease Management (Phone Group Counseling); PCMH (in clinic group visits) versus DM (phone group visits); Test type: Superiority; p = .025, Mixed Models Analysis; Mean Difference (Net) = -0.51, 97.5% CI 2-sided [-2.15 to 1.13]

2. Primary Outcome: Mean Weight Change Over 24 Months; Adjusted
Description: Mean weight change (kg) of participants between the three study groups. Weight loss at 24 months, and all relevant study visits in between, will be compared 1) between PCMH (in clinic group visits) versus FFS (in clinic individual visits), 2) between DM (phone group visits) versus FFS (in clinic individual visits), and 3) between PCMH (in clinic group visits) versus DM (phone group visits). Adjusted for affiliation, sex, race/ethnicity, education, diabetes, cardiovascular disease, and travel time to clinic.
Time Frame: Baseline and 6, 18 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (97.5% Confidence Interval); unit: kg
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
kg
  Mean weight change at 6 months | -6.01 [-7.72 to -4.31] | -8.62 [-10.23 to -7.00] | -7.97 [-9.63 to -6.32]
  Mean weight change at 18 months | -3.65 [-5.46 to -1.83] | -5.84 [-7.57 to -4.12] | -5.44 [-7.20 to -3.68]
  Mean weight change at 24 months | -2.85 [-4.67 to -1.03] | -4.69 [-6.42 to -2.96] | -4.19 [-5.96 to -2.42]
Statistical Analysis 1: Comparison: Fee-for-Service (In Clinic Individual Counseling) vs Patient Centered Medical Home (In Clinic Group Counseling); PCMH (in clinic group counseling) versus FFS (in clinic individual counseling); Test type: Superiority; p = .025, Mixed Models Analysis; Median Difference (Net) = -1.84, 97.5% CI 2-sided [-3.50 to -0.18]
Statistical Analysis 2: Comparison: Fee-for-Service (In Clinic Individual Counseling) vs Disease Management (Phone Group Counseling); DM (phone group counseling) versus FFS (in clinic individual counseling); Test type: Superiority; p = .025, Mixed Models Analysis; Median Difference (Net) = -1.34, 97.5% CI 2-sided [-2.99 to 0.32]
Statistical Analysis 3: Comparison: Patient Centered Medical Home (In Clinic Group Counseling) vs Disease Management (Phone Group Counseling); PCMH (in clinic group counseling) versus DM (phone group counseling); Test type: Superiority; p = .025, Mixed Models Analysis; Mean Difference (Net) = -0.50, 97.5% CI 2-sided [-2.15 to 1.15]

3. Secondary Outcome: Mean Percent Weight Loss Over 24 Months; Unadjusted Except for Affiliation
Description: Comparison in percent weight loss from baseline of participants between the three study groups. Weight loss at 24 months, and all relevant study visits in between, will be compared 1) between PCMH (in clinic group visits) versus FFS (in clinic individual visits), 2) between DM (phone group visits) versus FFS (in clinic individual visits), and 3) between PCMH (in clinic group visits) versus DM (phone group visits). Unadjusted except for affiliation.
Time Frame: Baseline and 6, 18 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: percentage from baseline
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
percentage from baseline
  Mean % weight change at 6 months | -5.58 [-6.49 to -4.68] | -8.20 [-9.08 to -7.32] | -7.52 [-8.41 to -6.63]
  Mean % weight change at 18 months | -3.23 [-4.27 to -2.19] | -5.47 [-6.49 to -4.46] | -5.06 [-6.09 to -4.03]
  Mean % weight change at 24 months | -2.48 [-3.53 to -1.43] | -4.30 [-5.33 to -3.27] | -3.83 [-4.87 to -2.79]

4. Secondary Outcome: Mean Change in Systolic Blood Pressure; Unadjusted Except for Affiliation
Description: Mean change in systolic blood pressure will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6, 18 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mmHg
  Mean change Systolic BP at 6 months | -2.41 [-4.57 to -0.25] | -2.08 [-4.19 to 0.03] | -2.27 [-4.39 to -0.15]
  Mean change Systolic BP at 18 months | -0.27 [-2.53 to 1.98] | -0.10 [-2.30 to 2.10] | -1.28 [-3.50 to 0.94]
  Mean change Systolic BP at 24 months | -0.58 [-2.80 to 1.63] | 0.12 [-2.05 to 2.28] | -1.60 [-3.77 to 0.58]

5. Secondary Outcome: Mean Change in Diastolic Blood Pressure; Unadjusted Except for Affiliation
Description: Mean change in diastolic blood pressure will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6, 18 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mmHg
  Mean change Diastolic BP at 6 months | -2.23 [-3.68 to -0.77] | -2.42 [-3.85 to -0.99] | -2.02 [-3.45 to -0.59]
  Mean change Diastolic BP at 18 months | -1.03 [-2.52 to 0.47] | -1.97 [-3.43 to -0.51] | -0.49 [-1.96 to 0.98]
  Mean change Diastolic BP at 24 months | -0.88 [-2.37 to 0.61] | -0.95 [-2.41 to 0.51] | -0.60 [-2.07 to 0.87]

6. Secondary Outcome: Mean Change in Fasting Glucose; Unadjusted Except for Affiliation
Description: Mean change in fasting glucose will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mg/dl
  Mean change fasting glucose at 6 months | -1.69 [-4.27 to 0.90] | -3.71 [-6.24 to -1.17] | -4.48 [-7.06 to -1.89]
  Mean change fasting glucose at 24 months | 3.07 [-0.07 to 6.21] | 0.94 [-2.17 to 4.04] | 0.29 [-2.88 to 3.47]

7. Secondary Outcome: Mean Change in Fasting Cholesterol; Unadjusted Except for Affiliation
Description: Mean change in fasting cholesterol will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mg/dl
  Mean change fasting cholesterol at 6 months | -6.20 [-9.52 to -2.87] | -8.22 [-11.48 to -4.96] | -5.89 [-9.21 to -2.56]
  Mean change fasting cholesterol at 24 months | -3.85 [-7.76 to 0.06] | -1.69 [-5.55 to 2.18] | -0.74 [-4.68 to 3.21]

8. Secondary Outcome: Mean Change in Fasting Triglycerides; Unadjusted Except for Affiliation
Description: Mean change in fasting triglycerides will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mg/dl
  Mean change fasting triglycerides at 6 months | -12.61 [-20.25 to -4.97] | -25.39 [-32.88 to -17.91] | -18.61 [-26.31 to -10.90]
  Mean change fasting triglycerides at 24 months | -0.46 [-8.22 to 7.30] | -19.17 [-26.78 to -11.56] | -10.40 [-18.23 to -2.57]

9. Secondary Outcome: Mean Change in Fasting Low Density Lipoprotein (LDL); Unadjusted Except for Affiliation
Description: Mean change in fasting low density lipoprotein (LDL) will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mg/dl
  Mean change fasting LDL at 6 months | -3.38 [-6.73 to -0.02] | -4.05 [-7.31 to -0.79] | -2.94 [-6.27 to 0.39]
  Mean change fasting LDL at 24 months | -5.26 [-9.13 to -1.39] | -1.38 [-5.17 to 2.41] | -0.83 [-4.72 to 3.05]

10. Secondary Outcome: Mean Change in Fasting High Density Lipoprotein (HDL); Unadjusted Except for Affiliation
Description: Mean change in fasting high density lipoprotein (HDL) will be compared across all treatment arms; unadjusted except for affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
mg/dl
  Mean change fasting HDL at 6 months | 0.25 [-1.27 to 1.77] | 0.76 [-0.73 to 2.24] | -0.05 [-1.56 to 1.46]
  Mean change fasting HDL at 24 months | 1.32 [-0.22 to 2.85] | 1.88 [0.38 to 3.39] | 2.12 [0.60 to 3.65]

11. Secondary Outcome: Mean Change in Physical Quality of Life Score, Measured by SF-12; Unadjusted Except for Affiliation
Description: Change in physical quality of life score, measured by SF-12. The Short Form Health Survey (SF-12) is a general quality of life measure with mental functioning and physical functioning summary scores. Each is scored from 0 to 100 with higher scores representing better functioning. Measures will be collected at baseline, 6 months and 24 months. Unadjusted Except for Affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
units on a scale
  Mean change SF-12 Physical Score at 6 months | 1.71 [0.83 to 2.59] | 2.69 [1.82 to 3.56] | 2.61 [1.72 to 3.49]
  Mean change SF-12 Physical Score at 24 months | 1.39 [0.43 to 2.34] | 1.50 [0.55 to 2.46] | 0.89 [-0.08 to 1.85]

12. Secondary Outcome: Mean Change in Mental Quality of Life Score, Measured by SF-12; Unadjusted Except for Affiliation
Description: Mean change in mental quality of life score, measured by SF-12. The Short Form Health Survey (SF-12) is a general quality of life measure with mental functioning and physical functioning summary scores. Each is scored from 0 to 100 with higher scores representing better functioning. Measures will be collected at baseline, 6 months and 24 months. Unadjusted Except for Affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
units on a scale
  Mean change SF-12 Mental Score at 6 months | 1.49 [0.35 to 2.64] | 1.92 [0.79 to 3.05] | -0.09 [-1.23 to 1.06]
  Mean change SF-12 Mental Score at 24 months | 0.89 [-0.28 to 2.05] | 0.93 [-0.22 to 2.09] | -0.07 [-1.24 to 1.10]

13. Secondary Outcome: Mean Change in Total Quality of Life Score Measured by IWQOL-L; Unadjusted Except for Affiliation
Description: The Impact of Weight on Quality of Life-Lite (IWQOL-L) measure consists of a total score and five subscales--physical function, self-esteem, sexual life, public distress, and work. The total score ranges from 0 to 100 with higher scores indicating better quality of life. Measures will be collected at baseline, 6 months and 24 months. Unadjusted Except for Affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
units on a scale
  Mean change IWQOL Total Score at 6 months | 11.16 [9.72 to 12.60] | 11.70 [10.28 to 13.11] | 11.73 [10.29 to 13.17]
  Mean change IWQOL Total Score at 24 months | 11.83 [10.23 to 13.42] | 11.32 [9.74 to 12.89] | 11.23 [9.63 to 12.83]

14. Secondary Outcome: Mean Change in Quality of Sleep Score Measured by PSQI; Unadjusted Except for Affiliation
Description: Measured using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 (better) to 21 (worse). Measures will be collected at baseline, 6 months and 24 months. Unadjusted Except for Affiliation.
Time Frame: Baseline and 6 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
units on a scale
  Mean Change PSQI Score at 6 months | -0.70 [-0.99 to -0.41] | -0.90 [-1.19 to -0.61] | -0.97 [-1.26 to -0.67]
  Mean Change PSQI Score at 24 months | -0.62 [-0.95 to -0.29] | -0.75 [-1.08 to -0.43] | -0.56 [-0.89 to -0.23]

15. Secondary Outcome: Mean Change in Stress Measured by PSS; Unadjusted Except for Affiliation
Description: Mean change in stress measured using the Perceived Stress Scale (PSS). Scores range from 0 to 40. Higher numbers represent greater levels of stress. Measures will be collected at baseline, 6 months, 18 months and 24 months. Unadjusted except for affiliation.
Time Frame: Baseline and 6, 18 and 24 months
Population: Enrolled minus deaths and medical removals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fee-for-Service (In Clinic Individual Counseling) | Patient Centered Medical Home (In Clinic Group Counseling) | Disease Management (Phone Group Counseling)
Number analyzed (Participants) | 473 | 468 | 466
units on a scale
  Mean change in PSS Score at 6 months | 0.03 [-0.39 to 0.46] | -0.33 [-0.75 to 0.09] | -0.26 [-0.68 to 0.17]
  Mean change in PSS Score at 18 months | 0.53 [0.11 to 0.96] | 0.46 [0.04 to 0.88] | 0.69 [0.26 to 1.12]
  Mean change in PSS Score at 24 months | -0.56 [-1.00 to -0.12] | -0.31 [-0.74 to 0.13] | -0.58 [-1.02 to -0.14]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs), to include deaths, were collected for each participant over an approximate two year period, from enrollment through the final study visit at 24 months.
Description: Only SAEs were captured for the study per approval of the overseeing Institutional Review Board (IRB) and the study Data Safety and Monitoring Board (DSMB). SAEs were identified during data collection visits at 6, 18 and 24 months, and via participant self-report surveys at 6, 12, 18 and 24 months. SAEs were also identified ad hoc via reporting by participants during study counseling sessions and during standard care clinic activities at each site.
Groups:
- Fee-for-Service (FFS; In Clinic Individual Counseling): Participants will receive individual counseling from their physician or other healthcare professional during regular clinic visits.
  Fee-for-Service Model (FFS): To be performed by participant's doctor or other healthcare professional in their doctor's office.
- Patient Centered Medical Home(PCMH;In Clinic Group Counseling): Participants will take part in group weight-management counseling during in-person group visits; later sessions may be conducted via group telephone calls if the group prefers.
  Patient Centered Medical Home (PCMH): To be performed by a registered dietitian, a nurse or other healthcare professional.
- Disease Management (DM; Phone Group Counseling): Participants will take part in group weight-management counseling by telephone.
  Disease Management (DM): To be performed by obesity treatment specialists with relevant graduate training and experience with weight loss counseling
Arm/Group | Fee-for-Service (FFS; In Clinic Individual Counseling) | Patient Centered Medical Home(PCMH;In Clinic Group Counseling) | Disease Management (DM; Phone Group Counseling)
All-Cause Mortality (participants affected / at risk) | 0/478 | 3/479 | 0/475
Serious Adverse Events (participants affected / at risk) | 94/478 | 88/479 | 82/475
Other Adverse Events (participants affected / at risk) | 0/478 | 0/479 | 0/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fee-for-Service (FFS; In Clinic Individual Counseling) (N=478) | Patient Centered Medical Home(PCMH;In Clinic Group Counseling) (N=479) | Disease Management (DM; Phone Group Counseling) (N=475)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Myelofibrosis, bone marrow transplant (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation with rapid ventricular response, ablation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest, secondary to ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain, cardiac, cardiac catheterization (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain, cardiac, myocardial infarction ruled out (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain, cardiac, unspecified EKG changes (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain, etiology unkown, myocardial infaction ruled out (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain, non-cardiac (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease, coronary artery bypass graft (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease, heart catheterizatrion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease, heart catheterizatrion, stent placement (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease, occluded stent, cardiac catheterization (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction, cardiac catheterization, stent placement (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction, coronary artery bypass graft (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction, Non-ST-elevation, cardiac catheterization (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia, supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congential scoliosis, broken rod, type unspecified, surgical repair (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Enlarged thyroid, benign, partial thyroidectomy (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism, total thyroidectomy (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Multinodular goiter, total thyroidectomy (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain, chronic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Clostridium difficile colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cystic fibrosis exacerbation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disesase (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Hernia, hiatal, surgical repair (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hernia, incisional, surgical repair (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hernia, inguinal, surgical repair (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia, umbilical, surgical repair (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hernia, unspecified, surgical repair (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea, vomiting, intractable (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Withdrawal reaction, acute, baclofen (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis, cholecysytectomy (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction, bee sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction, severe, etiology unspecified (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis, medication, not specified (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Medication reaction, IV contrast, chest pain (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis, exacerbation (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute febrile illness (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis, location not specified, post cat bile (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis, lower extermity (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis, mastectomy wound (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis, preauricular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis, upper extremity (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection, leg wound (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection, pacemaker (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection, pericarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection, periprosthetic, knee arthroplasty (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection, toe wound (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infection, urinary tract (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis, secondary to Group A strep infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis, secondary to influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis, secondary to pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis, secondary to urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration, severe (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Achilles tendon injury, surgical repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain, laminectomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bunion, bunionectomy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Charcot arthropathy, foot, surgical repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dislocation, internal hip prosthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture, ankle, surgical repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Fracture, humerus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture, knee, arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture, ribs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Injury, unspecifed, ankle, surgical repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Knee pain, arthroscopy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar degenerative disc disease, decompression surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lumbar degenerative disc disease, decompression, fusion surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis, cervical spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis, cervical spine, discectomy, fusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis, hip, arthoplasty (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 6 (6)
Osteoarthritis, knee, arthroplasty (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (11) | 9 (9)
Osteoarthritis, knee, arthroplasty revision (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis, knee, arthroplasty, bilateral (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Osteoarthritis, rotator cuff tear, shoulder, arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Osteomyelitis, ankle, surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis, shoulder, arthoplasty revision (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain, ankle, arthroplasty revision (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ruptured cervical vertebrae, surgical repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenomatoid nodule, partial thyroidectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer, lung, non-small cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer, prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer, prostate, prostatectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer, renal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer, thyroid, total thyroidectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Cancer, uterine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Gunshot wound, self-inflicted (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Pyleonephritis, acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure, acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal insufficency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal lithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic endocervicitis, paratubal cysts, hysterectomy, bilateral salpingo-oophorectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction, penile implant (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Fallopian tube torsion, surgical repair (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia, Hysterectomy (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1)
Menorrhagia, hysterectomy, recotocele repair (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic floor injury, hysterectomy, bladder sling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Post-hysterectomy prolapse, surgical repair (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease, exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Pneumonitis, interstitial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure, acute (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure, acute, secondary to bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure, acute, secondary to Influenza B (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsilitis, tonsillectomy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hemorrhage, post tonsillectomy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity Gastric Bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Capillary hemorrhage, leg (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 3 (3) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage, subarachnoid (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolus (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke-like symptoms (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope, near (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Syncope, recurrent (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attack (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Uncontrolled bleeding, post transurethral prostatectomy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT02456636/Prot_SAP_000.pdf